CLINICAL TRIAL: NCT00517413
Title: A Single-Arm Open-Label Study to Assess the Efficacy, Safety, and Tolerability of Once-Monthly Administration of Intravenous and/or Subcutaneous C.E.R.A for the Maintenance of Hemoglobin Levels in Dialysis Patients With Chronic Renal Anemia
Brief Title: LATINO Study: A Study of Mircera for the Maintenance Treatment of Dialysis Patients With Chronic Renal Anemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20881
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- C.E.R.A (Experimental): Participants with chronic renal anaemia who were on dialysis and previously treated with intravenous (IV) or subcutaneous (SC) epoetin alfa, epoetin beta or darbepoetin alfa received monthly treatment with Continuous Erythropoietin Receptor Activator (C.E.R.A.) (methoxy polyethylene glycol-epoetin beta [Mircera]). The initial dose of C.E.R.A. was based on the last dose of the previous Erythropoiesis Stimulating Agent (ESA); 120, 200, or 360 micrograms (mcg) C.E.R.A., IV or SC, every 4 weeks for 48 weeks.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 120, 200 or 360 micrograms sc or iv monthly, starting dose

SUMMARY:
This single arm study will assess the efficacy and safety of Mircera when administered once monthly, subcutaneously or intravenously, for the maintenance of hemoglobin levels in dialysis patients with chronic renal anemia. Patients currently receiving maintenance treatment with epoetin alfa will receive monthly injections of Mircera with a starting dose (120, 200 or 360 micrograms) derived from the dose of epoetin alfa they were receiving in the week preceding study start. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia;
* hemodialysis or peritoneal dialysis, with same mode of dialysis for >=3 months before and throughout screening period;
* stable maintenance epoetin alfa therapy for past 2 months.

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months;
* poorly controlled hypertension requiring interruption of epoetin alfa in past 6 months;
* acute or chronic bleeding during previous 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2007-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Santa Fe
- Brazil (4):
  - Aracajú
  - Curitiba
  - Fortaleza
  - São Paulo
- Santiago, Chile
- Bogotá, Colombia
- Quito, Ecuador
- Mexico (3):
  - Cuernavaca
  - Mexico City
  - Monterrey
- Peru (2):
  - Callao
  - Lima
- Montevideo, Uruguay
- Venezuela (2):
  - Caracas
  - Maracaibo

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 261 participants were screened and 163 participants were enrolled from 26 centers in 9 countries (Argentina, Brazil, Chile, Colombia, Ecuador, Mexico, Peru, Uruguay, Venezuela) from 08 October 2007 to 15 May 2010.
Period: Overall Study
Arm/Group | C.E.R.A
Started | 163
Completed | 102
Not Completed | 61
Not completed — Adverse Event | 7
Not completed — Death | 13
Not completed — Protocol Violation | 15
Not completed — Withdrawal by Subject | 2
Not completed — Failure to return | 1
Not completed — Other-Reasons | 23

BASELINE CHARACTERISTICS:
Population: The Intention To Treat (ITT) population included participants who received at least 1 dose of C.E.R.A. (Week 0) and for whom data for at least one follow-up variable were available.
Groups:
- C.E.R.A: Participants with chronic renal anaemia who were on dialysis and were previously treated with IV or SC epoetin alfa, epoetin beta or darbepoetin alfa, received monthly treatment with C.E.R.A. The initial dose of C.E.R.A. was based on the last dose of the previous ESA; 120, 200, or 360 mcg C.E.R.A., IV or SC, every 4 weeks for 48 weeks.
Arm/Group | C.E.R.A
Number analyzed (Participants) | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 94

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Their Mean Hb Concentration Within ±1.0 Gram/Deciliter of Their Reference Hb and Between 10.5 and 12.5 Gram/Deciliter
Description: The haemoglobin (Hb) levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The reference Hb value was defined on the basis of individual participant's all assessments at Weeks -4, -3, -2, -1 and 0. The Hb value on the first day of first dose (Week 0) was included in the calculation, as this assessment was performed before the first dose was given. The percentage of participants maintaining their mean Hb concentration within +/-1.0 gram/deciliter (g/dL) of their reference Hb and between 10.5 and 12.5 g/dL are reported for efficacy evaluation period (EEP). Efficacy evaluation period was from Week 16 to Week 24 after completion of 16-week dose titration period (DTP).
Time Frame: EEP (Week 16 to 24)
Population: The Per-Protocol Population (PP) included all participants in the safety population except those who had <3 recorded Hb values; withdrawn; inadequate iron defined as mean serum ferritin =<100 nanogram/milliliter (ng/mL) or mean TSAT=<20% or mean hypochromic RBCs>=10%; or had missing administration of C.E.R.A. all during EEP (Week 16-24).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 103
Percentage of participants | 43.7 [33.9 to 53.8]

2. Secondary Outcome: Mean Change in the Hb Concentration Between the Stability Verification Period and the EEP
Description: The Hb levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The mean change in the Hb concentration between the Stability Verification Period (SVP) and the EEP is reported.
Time Frame: SVP (Week -4 to -1), EEP (Week 16 to 24)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A
Number analyzed (Participants) | 161
g/dL | 0.08 (1.48)

3. Secondary Outcome: Percentage of Participants Maintaining Hb Concentration Within The Target Range 10.5 and 12.5 g/dL Throughout the EEP
Description: The Hb levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The percentage of participants maintaining their mean Hb concentration within the target range 10.5 and 12.5 g/dL throughout the EEP are reported.
Time Frame: EEP (Week 16 to 24)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 161
Percentage of participants | 47.8 [39.9 to 55.8]

4. Secondary Outcome: Mean Time Spent by the Participants in the Hb Target Range 10.5-12.5 g/dL During EEP
Description: The Hb levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The mean time (days) spent by the participants in the Hb target range 10.5 to 12.5 is reported.
Time Frame: EEP (Week 16 to 24)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: days
Arm/Group | C.E.R.A
Number analyzed (Participants) | 161
days | 30 (19.98)

5. Secondary Outcome: Mean C.E.R.A Dose To Maintain Hb Level Within the Range 10.5-12.5 g/dL Throughout the EEP
Description: The Hb levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The mean C.E.R.A dose required to maintain the Hb level within the range 10.5-12.5 g/dL throughout the EEP is presented.
Time Frame: EEP (Week 16 to 24)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | C.E.R.A
Number analyzed (Participants) | 161
mcg | 139.6 (86.58)

6. Secondary Outcome: Percentage of Participants Requiring Dose Adjustments of C.E.R.A During the DTP and EEP
Description: Dose adjustments were necessary when Hb increased or decreased by a clinically significant amount. The dose of C.E.R.A. was adjusted to maintain the individual participant's Hb within a range of +/-1.0 g/dL of the reference Hb concentration and between 10.5 and 12.5 g/dL throughout the DTP (Week 0 to Week 16) and the EEP (Weeks 16 to 24). The reference Hb value was taken as the mean of all Hb assessments during the stability verification period (Weeks -4, -3, -2, -1). The percentage of participants requiring C.E.R.A dose adjustments during the DTP and EEP are presented.
Time Frame: Baseline (Week 0) to Week 24
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 161
Percentage of participants
  Dose adjustment during DTP | 65.8
  Dose adjustment during EEP | 51.1

7. Secondary Outcome: Mean Monthly Dose of C.E.R.A During the DTP and EEP
Description: The initial dose of C.E.R.A. was 120, 200, or 360 mcg IV or SC every 4 weeks for 48 weeks, which was based on the last dose of the previous ESA. Dose adjustments were necessary when Hb increased or decreased by a clinically significant amount. The dose of C.E.R.A. was adjusted to maintain the individual participant's Hb within a range of +/-1.0 g/dL of the reference Hb concentration and between 10.5 and 12.5 g/dL throughout the DTP and the EEP. The reference Hb value was taken as the mean of all Hb assessments during the stability verification period. The mean monthly doses of C.E.R.A during the DTP and EEP are presented.
Time Frame: Baseline (Week 0) to Week 24
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | C.E.R.A
Number analyzed (Participants) | 161
mcg
  Mean monthly dose during DTP | 142.5 (50.32)
  Mean monthly dose during EEP | 139.6 (86.58)

8. Secondary Outcome: Incidence of Red Blood Cell Transfusions During the C.E.R.A. Treatment Phase
Description: Red blood cell (RBC) transfusions were permitted during the treatment period in case of medical need. The pre-transfusion Hb level was measured before any transfusion was administered.
Time Frame: Baseline (Week 0) to Week 44
Population: The safety population included all participants who entered into the study.
Measure: Number; unit: participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 162
participants | 13

9. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Adverse event (AE) and Serious adverse event (SAE) data was reported for the safety population which included all participants who entered into the study.
Time Frame: Up to Week 52
Population: The safety population included all participants who entered into the study.
Measure: Number; unit: participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 162
participants
  Participants with AE | 120
  Participants with SAE | 53

10. Secondary Outcome: Mean Haemoglobin Levels Over Time
Description: The Hb levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The standard reference range for Hb are as follows: Female: min-max for lower limit=11 to 13 g/dL and min-max for upper limit=14 to 18.1 g/dL; Male: min-max for lower limit=12 to 14.2 g/dL and min-max for upper limit=16 to 18.1 g/dL.
Time Frame: Baseline (Week 0), Week 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: The safety population included all participants who entered into the study. n = the number of participants analyzed at a given time point.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A
Number analyzed (Participants) | 162
g/dL
  Hb at Week 0 (n=162) | 11.4 (0.58)
  Hb at Week 8 (n=151) | 11.7 (1.44)
  Hb at Week 12 (n=144) | 11.7 (1.67)
  Hb at Week 16 (n=141) | 11.6 (1.56)
  Hb at Week 20 (n=137) | 11.5 (1.65)
  Hb at Week 24 (n=132) | 11.6 (1.36)
  Hb at Week 28 (n=121) | 11.8 (1.38)
  Hb at Week 32 (n=120) | 11.6 (1.62)
  Hb at Week 36 (n= 114) | 11.7 (1.58)
  Hb at Week 40 (n=110) | 11.7 (1.31)
  Hb at Week 44 (n=105) | 11.5 (1.39)
  Hb at Week 48 (n=103) | 11.4 (1.27)

11. Secondary Outcome: Mean Hematocrit Levels Over Time
Description: The haematocrit (HCT) levels in fraction were recorded for each participant at enrollment and at different time points during the study up to Week 48. The standard reference range for hematocrit are as follows: Female: min-max for lower limit=0.12 - 0.38 and min-max of upper limit=0.43 - 0.537; Male: min-max for lower limit=0.35 - 0.45 and min-max of upper limit=0.45 - 0.54.
Time Frame: Baseline (Week 0), Week 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | C.E.R.A
Number analyzed (Participants) | 162
Proportion of red blood cells in blood
  HCT at Week 0 (n=162) | 0.35 (0.02)
  HCT at Week 8 (n=151) | 0.35 (0.05)
  HCT at Week 12 (n=139) | 0.36 (0.05)
  HCT at Week 16 (n=141) | 0.35 (0.05)
  HCT at Week 20 (n=132) | 0.35 (0.05)
  HCT at Week 24 (n=132) | 0.35 (0.04)
  HCT at Week 28 (n=117) | 0.36 (0.04)
  HCT at Week 32 (n=119) | 0.36 (0.05)
  HCT at Week 36 (n=110) | 0.36 (0.05)
  HCT at Week 40 (n=110) | 0.36 (0.04)
  HCT at Week 44 (n=101) | 0.35 (0.04)
  HCT at Week 48 (n=103) | 0.35 (0.04)

12. Secondary Outcome: Mean White Blood Cells and Thrombocyte Levels Over Time
Description: The white blood cells (WBC) and thrombocyte levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The standard reference ranges for WBC are as follows: Female/Male: min-max for lower limit= 3.5 - 5*10^9 cells/L and min-max of upper limit= 9 -13.5*10^9 cells/L. The standard reference ranges for thrombocyte are as follows: Female/Male: min-max for lower limit= 130 - 150*10^9 cells/L and min-max of upper limit= 300 - 450*10^9 cells/L.
Time Frame: Baseline (Week 0), Week 8, 16, 24, 32, 40, and 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 160
10^9 cells/L
  WBC at Week 0 (n=160) | 6.8 (1.90)
  WBC at Week 8 (n=147) | 6.5 (2.10)
  WBC at Week 16 (n=137) | 6.7 (2.01)
  WBC at Week 24 (n=130) | 6.6 (2.09)
  WBC at Week 32 (n=116) | 6.6 (1.78)
  WBC at Week 40 (n=106) | 6.6 (2.19)
  WBC at Week 48 (n=101) | 6.6 (1.98)
  Thrombocyte at Week 0 (n=159) | 219.7 (59.73)
  Thrombocyte at Week 8 (n=144) | 204.4 (56.21)
  Thrombocyte at Week 16 (n=135) | 207.4 (57.76)
  Thrombocyte at Week 24 (n=129) | 205.2 (52.28)
  Thrombocyte at Week 32 (n=117) | 207.9 (69.97)
  Thrombocyte at Week 40 (n=105) | 209.3 (55.95)
  Thrombocyte at Week 48 (n=101) | 209.0 (58.38)

13. Secondary Outcome: Mean Phosphate and Potassium Levels Over Time
Description: The phosphate and potassium levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The standard reference ranges for phosphate are as follows: Female/Male: min-max for lower limit= 0.48435 - 0.9687 mmol/L and min-max for upper limit=1.45305 - 2.2603 mmol/L. The standard reference ranges for potassium are as follows: Female/Male: min-max for lower limit=3.1 - 3.7 mmol/L and min-max for upper limit=5 - 5.5 mmol/L.
Time Frame: Baseline (Week 0), Week 8, 16, 24, 32, 40, and 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 159
mmol/L
  Phosphate at Week 0 (n=154) | 1.61 (0.55)
  Phosphate at Week 8 (n=135) | 1.69 (0.59)
  Phosphate at Week 16 (n=131) | 1.70 (0.57)
  Phosphate at Week 24 (n=125) | 1.68 (0.57)
  Phosphate at Week 32 (n=110) | 1.60 (0.61)
  Phosphate at Week 40 (n=105) | 1.59 (0.60)
  Phosphate at Week 48 (n=97) | 1.61 (0.65)
  Potassium at Week 0 (n=159) | 4.90 (0.87)
  Potassium at Week 8 (n=133) | 4.80 (0.86)
  Potassium at Week 16 (n=133) | 4.90 (0.87)
  Potassium at Week 24 (n=124) | 4.90 (0.89)
  Potassium at Week 32 (n=110) | 4.80 (0.83)
  Potassium at Week 40 (n=104) | 4.80 (0.88)
  Potassium at Week 48 (n=99) | 5.00 (0.90)

14. Secondary Outcome: Mean Creatinine, Iron, and Total Iron Binding Capacity Levels Over Time
Description: The creatinine, iron, and total iron binding capacity (TIBC) levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The standard reference ranges for creatinine are as follows: Female: min-max for lower limit=0 - 70.72 mmol/L and min-max for upper limit=79.56 - 123.76 mmol/L; Male: min-max for lower limit=0 - 70.72 mmol/L and min-max for upper limit=97.24 - 123.76 mmol/L. The standard reference ranges for iron are as follows: Female: min-max for lower limit=6.265 - 10.74 mmol/L and min-max for upper limit=25.06 - 32.22 mmol/L and Male: min-max for lower limit=6.265 - 11.635 mmol/L and min-max for upper limit=25.06 - 32.22 mmol/L. The standard reference ranges for TIBC are as follows: Female: min-max for lower limit=19.69 - 49.046 mmol/L and min-max for upper limit=62.65 - 88.963 mmol/L and Male: min-max for lower limit=19.69 - 52.089 mmol/L and min-max for upper limit=62.65 - 80.55 mmol/L.
Time Frame: Baseline (Week 0), Week 8, 16, 24, 32, 40, and 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 159
μmol/L
  Creatinine at Week 0 (n=153) | 847.1 (269.15)
  Creatinine at Week 8 (n=120) | 823.4 (274.17)
  Creatinine at Week 16 (n=122) | 814.0 (268.76)
  Creatinine at Week 24 (n=118) | 822.9 (265.76)
  Creatinine at Week 32 (n=112) | 804.5 (284.33)
  Creatinine at Week 40 (n=95) | 809.7 (292.23)
  Creatinine at Week 48 (n=93) | 816.6 (315.21)
  Iron at Week 0 (n=159) | 13.9 (6.28)
  Iron at Week 8 (n=136) | 16.0 (6.79)
  Iron at Week 16 (n=133) | 17.6 (9.79)
  Iron at Week 24 (n=121) | 16.5 (8.12)
  Iron at Week 32 (n=110) | 16.0 (8.28)
  Iron at Week 40 (n=99) | 16.3 (7.75)
  Iron at Week 48 (n=97) | 14.4 (6.55)
  TIBC at Week 0 (n=97) | 38.5 (10.38)
  TIBC at Week 8 (n=75) | 39.7 (11.23)
  TIBC at Week 16 (n=74) | 41.5 (11.99)
  TIBC at Week 24 (n=76) | 42.0 (19.80)
  TIBC at Week 32 (n=68) | 41.4 (11.97)
  TIBC at Week 40 (n=66) | 39.6 (9.31)
  TIBC at Week 48 (n=58) | 44.0 (23.57)

15. Secondary Outcome: Mean Transferrin Saturation Levels Over Time
Description: Transferrin saturation (TSAT) is the ratio of serum iron and total iron-binding capacity. Transferrin is a blood protein that picks up iron absorbed by the intestines and transports it from one location to another. When iron absorption is abnormally high, transferrin proteins become more saturated with iron. An elevated TS value therefore reflects an increase in iron absorption. The TSAT levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. TSAT was calculated automatically in the electronic case report form (eCRF) according to the following formulae: TSAT= (Serum Iron*100)/(Transferrin*1.41) or TSAT=(Serum Iron*100)/TIBC. Calculated data was not provided by laboratory; therefore no reference range is available.
Time Frame: Baseline (Week 0), Week 8, 16, 24, 32, 40, and 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of Transferrin Saturation
Arm/Group | C.E.R.A
Number analyzed (Participants) | 135
Percentage of Transferrin Saturation
  TSAT at Week 0 (n=135) | 34.7 (19.16)
  TSAT at Week 8 (n=113) | 39.8 (19.52)
  TSAT at Week 16 (n=113) | 46.3 (28.26)
  TSAT at Week 24 (n=108) | 42.1 (22.20)
  TSAT at Week 32 (n=96) | 39.3 (24.83)
  TSAT at Week 40 (n=91) | 40.2 (21.85)
  TSAT at Week 48 (n=84) | 36.8 (21.56)

16. Secondary Outcome: Mean Albumin and Transferrin Levels Over Time
Description: The albumin and transferrin levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The standard reference ranges for albumin are as follows: Female/Male: min-max for lower limit=30 - 35 g/L and min-max for upper limit=48 - 55 g/L. The standard reference ranges for transferrin are as follows: Female/Male: min-max for lower limit=1.5 - 2.3 g/L and min-max for upper limit=2.87 - 4.3 g/L.
Time Frame: Baseline (Week 0), Week 8, 16, 24, 32, 40, and 48
Population: The safety population included all participants who entered into the study.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 157
g/L
  Albumin at Week 0 (n=157) | 39.5 (4.61)
  Albumin at Week 8 (n=134) | 39.3 (5.10)
  Albumin at Week 16 (n=134) | 39.3 (5.96)
  Albumin at Week 24 (n=124) | 39.3 (5.40)
  Albumin at Week 32 (n=111) | 39.4 (6.24)
  Albumin at Week 40 (n=99) | 39.9 (5.25)
  Albumin at Week 48 (n=98) | 39.6 (4.96)
  Transferrin at Week 0 (n=75) | 1.82 (0.47)
  Transferrin at Week 8 (n=57) | 1.84 (0.54)
  Transferrin at Week 16 (n=63) | 1.81 (0.54)
  Transferrin at Week 24 (n=54) | 1.90 (0.49)
  Transferrin at Week 32 (n==44) | 1.91 (0.60)
  Transferrin at Week 40 (n=47) | 1.96 (0.59)
  Transferrin at Week 48 (n=46) | 2.96 (7.48)

17. Secondary Outcome: Mean C-Reactive Protein Levels Over Time
Description: C-reactive protein (CRP) is produced by the liver. The level of CRP rises when there is inflammation throughout the body. The CRP test is a general test to check for inflammation in the body.The CRP levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The standard reference ranges for CRP are as follows: Female/Male: min-max for lower limit=0 - 10 mg/L and min-max for upper limit=0.5 - 30 mg/L.
Time Frame: Baseline (Week 0), 8, 16, 24, 32, 40, and 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 113
mg/L
  CRP at Week 0 (n=113) | 54.1 (147.89)
  CRP at Week 8 (n=102) | 87.5 (218.41)
  CRP at Week 16 (n=107) | 186.8 (1414.66)
  CRP at Week 24 (n=104) | 64.0 (163.67)
  CRP at Week 32 (n=94) | 53.4 (118.21)
  CRP at Week 40 (n=84) | 250.6 (1890.84)
  CRP at Week 48 (n=88) | 61.7 (169.60)

18. Secondary Outcome: Mean Ferritin Levels Over Time
Description: Ferritin is a protein found inside cells that stores iron so that the body can use it later. A ferritin test indirectly measures the amount of iron in your blood. The Ferritin levels were recorded for each participant at enrollment and at different time points during the study up to Week 48. The standard reference ranges for ferritin are as follows: Female: min-max for lower limit=6 - 50 mcg/L and min-max for upper limit=120 - 400 mcg/L; Male: min-max for lower limit=10 - 50 mcg/L and min-max for upper limit=200 - 400 mcg/L.
Time Frame: Baseline (Week 0), Week 8, 16, 24, 32, 40, and 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 157
mcg/L
  Ferritin at Week 0 (n=157) | 591.8 (420.67)
  Ferritin at Week 8 (n=134) | 617.0 (428.36)
  Ferritin at Week 16 (n=131) | 598.8 (408.20)
  Ferritin at Week 24 (n=123) | 578.5 (403.87)
  Ferritin at Week 32 (n=110) | 583.0 (478.92)
  Ferritin at Week 40 (n=98) | 591.2 (457.24)
  Ferritin at Week 48 (n=97) | 590.3 (433.97)

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: Adverse event (AE) and Serious adverse event (SAE) data was reported for the safety population which included all participants who entered into the study.
Arm/Group | C.E.R.A
Serious Adverse Events (participants affected / at risk) | 53/162
Other Adverse Events (participants affected / at risk) | 40/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A (N=162)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina Pectoris (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Cardiogenic Shock (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Adrenal Insufficiency (Endocrine disorders) | 1
Visual Acuity Reduced (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum Intestinal (Gastrointestinal disorders) | 1
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1
Gastritis Erosive (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3
Haematemesis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Inguinal Hernia (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Sudden death (General disorders) | 2
Cellulitis (Infections and infestations) | 1
Device Related Infection (Infections and infestations) | 1
Device Related Sepsis (Infections and infestations) | 1
Diabetic Foot Infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Muscle Abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Respiratory Tract Infection (Infections and infestations) | 1
Septic Shock (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 5
Face Injury (Injury, poisoning and procedural complications) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1
Vascular Access Complication (Injury, poisoning and procedural complications) | 1
Vascular Bypass Dysfunction (Injury, poisoning and procedural complications) | 1
Haemoglobin Decreased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Paraneoplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Vascular Dementia (Nervous system disorders) | 1
Vascular Headache (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1
Renal Transplant (Surgical and medical procedures) | 1
Aortic Dissection (Vascular disorders) | 1
Arterial Thrombosis Limb (Vascular disorders) | 1
Extremity Necrosis (Vascular disorders) | 1
Hypertensive Crisis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Peripheral Ischaemia (Vascular disorders) | 1
Shock Haemorrhagic (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Venous Stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A (N=162)
Diarrhoea (Gastrointestinal disorders) | 11
Hypertension (Vascular disorders) | 24
Hypotension (Vascular disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.